CLINICAL TRIAL: NCT04860973
Title: A Feasibility Study of Weighted Blankets to Help Agitation and Disturbed Sleep After Brain Injury
Brief Title: Weighted Blankets After Brain Injury
Acronym: WEBLY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Of those randomised to intervention arm, the majority were not able to tolerate the intervention for the duration of the study indicating that it is not feasible on a larger scale and recruiting 2 extra participants would not change this decision.
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHDB/2020/024
Record Dates: First submitted 2020-09-08; First posted 2021-04-27 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weighted blankets (Experimental): Provided with weighted blanket suitable for participant's weight
  Interventions: Device: Weighted blankets
- Standard linen (No Intervention): Use of standard hospital linen

INTERVENTIONS:
Device: Weighted blankets — Weighted blankets given to patient for 7 days/nights
  Arms: Weighted blankets

SUMMARY:
A non-blinded randomised controlled feasibility study of weighted blankets to help agitation and disturbed sleep after brain injury. This is a single centre study based in a community hospital in the UK. Outcomes centre on determining the feasibility and acceptability of the study taking place in an NHS setting.

DETAILED DESCRIPTION:
A non-blinded randomised controlled feasibility study of weighted blankets to help agitation and disturbed sleep after brain injury. This is a single centre study based in a community hospital in the UK. Outcomes centre on determining the feasibility and acceptability of the study taking place in an NHS setting.

12 subjects will be randomised 1:1 to intervention or control; they will use the allocated linen for 7 consecutive days and nights. Sleep will be measured using observations and actigraphs; behaviour and behavioural interventions will be recorded.

Participants (where possible) and staff members will be interviewed about their experience and opinions.

ELIGIBILITY:
Inclusion Criteria

* Subjects capable of giving informed consent, or if appropriate, subjects having an acceptable individual capable of giving assent on the subject's behalf
* Aged over 18 years
* Admitted to King's Lodge Neurorehabilitation Unit for inpatient rehabilitation after a brain injury
* Within weight limits to be suitable for weighted blanket use

Exclusion Criteria

* On end of life pathway
* Pain which could be exacerbated by weighted blanket
* Unable to remove
* Presence of open wound / pressure sore
* Allergy to blanket material
* Participant or consultee unable or unwilling to give informed consent / assent
* Known respiratory disorder such as asthma, chronic obstructive pulmonary disease, obstructive sleep apnoea which could be exacerbated by use of heavy blanket over chest
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Recruitment | 12 months
  Proportion of eligible candidates recruited within the time frame

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Derby & Burton NHS Foundation Trust, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No